CLINICAL TRIAL: NCT07193251
Title: The Effects of Connective Tissue Massage Combined With Core Stabilization Exercises on Pain, Functionality, and Endurance in Mechanical Low Back Pain
Brief Title: Connective Tissue Massage and Core Training in Mechanical Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Burcu AKKURT, PhD, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1234
Record Dates: First submitted 2025-09-18; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Mechanical Low Back Pain
Keywords: mechanical low back pain; connective tissue massage; core stabilization exercise
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core stabilization+connective tissue massage (Experimental): Participants will receive supervised core stabilization exercises twice weekly for 8 weeks (≈50 min: 10 min warm-up, 30 min stabilization, 10 min cool-down), progressing from basic trunk activation and bridging to plank and ball-assisted tasks. A daily 60-min home program with illustrated handouts will be prescribed. In addition, each supervised session will include 20 min of connective tissue massage (CTM) applied bilaterally to lumbar and lower thoracic regions using oblique and transverse pulls at connective tissue reflex zones. CTM will be performed in seated or prone position depending on patient comfort. Interventions will be delivered under physiotherapist supervision in the university physiotherapy laboratories.
  Interventions: Other: Core Stabilization Exercises; Other: Connective tissue massage
- Core Stabilization Exercises Only (Active Comparator): Participants will receive the same supervised core stabilization program as the experimental arm (twice weekly for 8 weeks, ≈50 min per session with progressive exercises from activation to advanced tasks) and the same daily 60-min home exercise prescription. No connective tissue massage will be provided. Sessions will be delivered under physiotherapist supervision in the same laboratory setting to ensure consistency across arms.
  Interventions: Other: Core Stabilization Exercises

INTERVENTIONS:
Other: Core Stabilization Exercises — Participants will receive supervised core stabilization exercises twice weekly for 8 weeks (≈50 min: 10 min warm-up, 30 min stabilization, 10 min cool-down), progressing from basic trunk activation and bridging to plank and ball-assisted tasks. A daily 60-min home program with illustrated handouts will be prescribed.
Other: Connective tissue massage — each supervised session will include 20 min of connective tissue massage (CTM) applied bilaterally to lumbar and lower thoracic regions using oblique and transverse pulls at connective tissue reflex zones. CTM will be performed in seated or prone position depending on patient comfort
  Arms: Core stabilization+connective tissue massage

SUMMARY:
This randomized controlled study will investigate the effects of connective tissue massage combined with core stabilization exercises in patients with mechanical low back pain. Participants will be assigned to two groups: one will receive core stabilization exercises with connective tissue massage, while the other will receive only core stabilization exercises. Pain will be evaluated using the Visual Analog Scale, functionality will be assessed with the Oswestry Disability Index, and endurance will be measured with static and dynamic curl-up, static back endurance, and side bridge tests. Quality of life will be assessed with the SF-36, and instrumental daily living activities will be evaluated with the Lawton & Brody Scale. The results will demonstrate whether adding connective tissue massage to core stabilization exercises will provide additional benefits in pain reduction, functional improvement, endurance, and quality of life compared to exercises alone.

DETAILED DESCRIPTION:
This randomized controlled clinical trial will evaluate the effects of connective tissue massage (CTM) combined with core stabilization exercises (CSEs) on pain, functionality, endurance, and quality of life in patients with mechanical low back pain. A total of 29-30 participants aged 20 to 55 years who will be diagnosed with mechanical low back pain will be recruited. Participants will be randomized into two groups:

Experimental group: will receive core stabilization exercises plus connective tissue massage.

Control group: will receive only core stabilization exercises.

All interventions will be delivered under physiotherapist supervision in the physiotherapy and rehabilitation laboratories. The exercise program will include progressive core stabilization exercises performed twice per week for eight weeks, each session lasting approximately 50 minutes (10 minutes warm-up, 30 minutes core stabilization, 10 minutes cool-down). The experimental group will additionally receive 20 minutes of connective tissue massage twice per week during the same 8-week intervention period.

Outcome measures will include:

Pain: Visual Analog Scale (VAS).

Functionality: Oswestry Disability Index.

Endurance: Static and dynamic curl-up, static back endurance, and horizontal side bridge tests.

Lumbar mobility: Finger-to-floor distance.

Muscle strength: Manual muscle testing.

Quality of life: Short Form-36 (SF-36).

Instrumental activities of daily living: Lawton & Brody Instrumental ADL Scale.

Assessments will be performed at baseline and after the 8-week intervention period. The study will hypothesize that connective tissue massage combined with core stabilization exercises will provide greater improvements in pain relief, functional status, muscular endurance, and quality of life compared to core stabilization exercises alone.

The results will contribute evidence on whether connective tissue massage will offer an additional therapeutic benefit when integrated into a rehabilitation program for patients with mechanical low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be 20-55 years of age.
* Participants will have a clinician-confirmed diagnosis of mechanical low back pain and will be referred by specialists in Physical Medicine and Rehabilitation.
* Participants will have adequate cognitive ability to follow assessments and the treatment protocol and will agree to attend supervised sessions (2×/week for 8 weeks) and to perform daily home exercises.
* Participants will provide informed consent prior to any study procedures

Exclusion Criteria:

* Participants will be excluded if they have a history of lumbar spine surgery.
* Participants will be excluded for conditions affecting the lumbar region, including inflammatory arthritis, tumor, or infectious diseases.
* Participants will be excluded if they present congenital anomalies of the lumbosacral region or secondary orthopedic problems that could interfere with the study.
* Participants will be excluded if they have neurological disorders (e.g.,Parkinson's disease, Alzheimer's disease, multiple sclerosis) or systemic diseases such as diabetes mellitus.
* Any medical condition judged by the investigators to preclude safe participation or adherence to the protocol will lead to exclusion.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | From enrollment to the end of treatment at 8 weeks
  Functional status will be assessed with the ODI, a 10-item questionnaire scored from 0 to 5 per item, covering pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, traveling, and changing pain intensity. Scores will be converted into percentages, with higher scores indicating greater disability. The total score will be calculated as a percentage, where 0% indicates no disability and 100% represents the highest level of disability.
Visual Analog Scale (VAS) | From enrollment to the end of treatment at 8 weeks
  Pain intensity will be measured using the Visual Analog Scale, a 10-cm horizontal line ranging from 0 ("no pain") to 10 ("worst pain imaginable"). Higher scores will indicate greater pain severity.
Curl-Up Test (Static and Dynamic) | From enrollment to the end of treatment at 8 weeks
  Abdominal endurance will be measured by static and dynamic curl-up tests. For the static test, participants will maintain a standardized trunk-flexion position until fatigue. For the dynamic test, participants will perform as many curl-ups as possible within 1 minute. Longer holding times or higher repetitions will indicate greater endurance. Measured in seconds/repetitions, with higher values indicating greater endurance.
Biering-Sørensen Test | From enrollment to the end of treatment at 8 weeks.
  Back extensor endurance will be evaluated by maintaining the upper body in a horizontal position over the edge of a table while the pelvis and legs are stabilized. Time will be recorded in seconds, with longer duration indicating greater endurance. Higher scores will indicate greater endurance.
Side Bridge Test | From enrollment to the end of treatment at 8 weeks.
  Spinal stabilizer endurance will be measured in a side-lying position with support on the elbow and feet. Participants will elevate the pelvis to align the body horizontally and maintain this position as long as possible. Longer holding times will indicate higher endurance capacity. The test will be terminated when the participant can no longer maintain the straight body position or after 240 seconds. Higher scores will indicate greater endurance.

SECONDARY OUTCOMES:
Finger-to-Floor Distance Test | From enrollment to the end of treatment at 8 weeks
  Lumbar spine flexibility will be assessed by asking participants to bend forward with knees extended and attempt to touch the floor. The distance in centimeters between the fingertips and the floor will be measured. Smaller distances will indicate better mobility.
Manual Muscle Testing (MMT, Lovett Scale) | From enrollment to the end of treatment at 8 weeks
  Flexibility of hip flexors, hamstrings, and lumbar extensors will be assessed through standardized muscle length tests. Presence of limited range will indicate muscle tightness.
Short Form-36 Health Survey (SF-36) | From enrollment to the end of treatment at 8 weeks
  Health-related quality of life will be evaluated using the SF-36, consisting of 8 subscales (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, mental health). Each domain is scored from 0 to 100, with higher scores reflecting better health status.
Lawton & Brody Instrumental Activities of Daily Living (IADL) Scale | From enrollment to the end of treatment at 8 weeks
  Functional independence in daily living will be assessed with the IADL scale, which includes activities such as using the telephone, shopping, food preparation, housekeeping, laundry, transportation, medication management, and handling finances. Scores range from 0 to 24, with higher scores indicating greater independence.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No